CLINICAL TRIAL: NCT00360724
Title: Duloxetine for Chronic Depression: a Double-blind Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: # 4967/6363R
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Dysthymic Disorder; Depressive Disorder NOS
Keywords: dysthymia; dysthymic disorder; chronic depression; chronic low-grade depression; atypical depression; minor depression; depression NOS; depression; depressive disorder; mood disorder; unipolar depression; low-grade depression
MeSH Terms: conditions — Dysthymic Disorder; Depression; Depressive Disorder; Mood Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- duloxetine (cymbalta) (Experimental): Duloxetine medication: a medication currently marketed in the USA that is reported to have pharmacological effects including reuptake blockage for serotonin and norepinephrine
  Interventions: Drug: Duloxetine (Cymbalta)
- Placebo treatment (Placebo Comparator): placebo treatment: treatment with placebo capsules that match active medication capsules
  Interventions: Drug: Duloxetine (Cymbalta)

INTERVENTIONS:
Drug: Duloxetine (Cymbalta) — duloxetine medication up to dose of 120 mg/day
  Other Names: duloxetine; Cymbalta

SUMMARY:
The investigators are studying a new antidepressant medicine, duloxetine, for the treatment of people with chronic depression. Duloxetine (trade name Cymbalta) was recently approved by the FDA for the treatment of major depression. The investigators are testing whether this medicine is also effective for adults with chronic depression (dysthymic disorder or dysthymia).

Chronic depression, lasting two or more years, often causes significant suffering and impairment. The investigators study involves a 6 to 10 week double-blind Initial Phase during which half of the participants will take the new medication and half will take a placebo (an inactive look-alike pill). After the Initial Phase, a 12-week Continuation Phase will begin, during which all subjects can be treated with an FDA-approved antidepressant medication.

Eligible subjects may also receive MRI scans, to help the investigators understand how antidepressants work in treating depression.

DETAILED DESCRIPTION:
This is a 22-week study of the tolerability, dosing, and efficacy of duloxetine in chronically depressed outpatients. Participants can have Dysthymic Disorder (Dysthymia), or Depression, Not Otherwise Specified (Depression NOS).

The first 10 weeks (Acute Phase) are double blind, placebo-controlled, and the second 12 weeks (Continuation Phase) is open-label and all subjects will receive active medication.

Tests of cytokine functioning will be performed and analyzed for treatment and placebo effects.

In addition, a subset of patients will be enrolled into an Magnetic Resonance Imaging (MRI) sub-study, in which a variety of brain imaging techniques (including anatomical MRI, functional MRI (fMRI), MR Spectroscopy, and Diffusion Tensor Imaging) will be performed at baseline and week 10. Duloxetine responders will have a third MRI performed at week 22.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 75 years (ages 20 to 60 for MRI sub-study)
* diagnosis of dysthymic disorder (chronic depression) or depression NOS
* minimum of 2 years duration of current episode of depression

Exclusion Criteria:

* current major depression
* diagnoses including delirium, dementia, bipolar disorder, schizophrenia
* substance abuse or dependence in the past 6 months
* pregnant or nursing women
* serious risk of suicide

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Hellerstein, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hellerstein DJ, Stewart JW, McGrath PJ, Deliyannides DA, Batchelder ST, Black SR, Withers A, O'Shea D, Chen Y. A randomized controlled trial of duloxetine versus placebo in the treatment of nonmajor chronic depression. J Clin Psychiatry. 2012 Jul;73(7):984-91. doi: 10.4088/JCP.11m07230. PMID 22901348
- [Derived] Yang J, Hellerstein DJ, Chen Y, McGrath PJ, Stewart JW, Peterson BS, Wang Z. Serotonin-norepinephrine reuptake inhibitor antidepressant effects on regional connectivity of the thalamus in persistent depressive disorder: evidence from two randomized, double-blind, placebo-controlled clinical trials. Brain Commun. 2022 Apr 15;4(3):fcac100. doi: 10.1093/braincomms/fcac100. eCollection 2022. PMID 35592490
- [Derived] Bansal R, Hellerstein DJ, Sawardekar S, O'Neill J, Peterson BS. Effects of the antidepressant medication duloxetine on brain metabolites in persistent depressive disorder: A randomized, controlled trial. PLoS One. 2019 Jul 19;14(7):e0219679. doi: 10.1371/journal.pone.0219679. eCollection 2019. PMID 31323045
- [Derived] Hellerstein DJ, Hunnicutt-Ferguson K, Stewart JW, McGrath PJ, Keller S, Peterson BS, Chen Y. Do social functioning and symptoms improve with continuation antidepressant treatment of persistent depressive disorder? An observational study. J Affect Disord. 2017 Mar 1;210:258-264. doi: 10.1016/j.jad.2016.12.026. Epub 2016 Dec 20. PMID 28064115
- See also: Mood Disorders Research Program website — http://www.DepressionNY.com
- See also: Columbia University Department of Psychiatry website — http://asp.cumc.columbia.edu/facdb/psychiatry/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by advertisements, website postings, and from the hospital's telephone referral service. Conducted between August 2006 and December 2011. Potential participants provided informed consent for study participation. A physical examination was performed and blood and urine samples were collected, including urine toxicology.
Pre-assignment Details: For patients on current ineffective psychotropic medication, washout was required, with >=7 days medication-free (>=28 days for fluoxetine). Concurrent sleep medication (zolpidem) was allowed for a maximum of 5 days during the study.
Groups:
- Duloxetine (Cymbalta): Duloxetine medication, ranging from 30 to 120 mg/day
- Placebo Treatment: placebo treatment, treatment with matching capsules of placebo
Period: Overall Study
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Started | 33 | 32
Completed | 29 | 28
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.7) | 42.1 (11.4) | 41.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 15 | 22 | 37
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS) - 24 Total Score
Description: HDRS-24 total score, standardly used rating scale for depression. Score 0-7 no depression; Score 8-16 mild depression; Score 17-23 moderate depression; Score 24 and up severe depression. Range= 0 to 75, higher score=worse depression
Time Frame: Week 10
Population: Patients for whom post-baseline data was available and scored 2 or less on the suicide item either at baseline or during the course of treatment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo Treatment: placebo treatment, with capsules matching the duloxetine medication
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
Scores on a scale | 5 (3.6) | 10 (5.5)
Statistical Analysis 1: Comparison: Duloxetine (Cymbalta) vs Placebo Treatment; Repeated measures ANOVA was used to compare measures between baseline and week 10; Test type: Superiority or Other; p = .003, Repeated Measures ANOVA; df 1,55; F statistics = 9.43 — time X Drug group, f=9.43,df 1,55, p=.003

2. Primary Outcome: Hamilton Depression Rating Scale (HDRS) - 24 Total Score
Description: as for outcome 1
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
Scores on a scale | 14.1 (3.8) | 14.9 (3.5)

3. Secondary Outcome: Cornell Dysthymia Rating Scale (CDRS)
Description: CDRS is a 20-item clinician-rated inventory for chronic depressive symptoms. Each item was characterized by an explanatory or illustrative description and rated from 0 (symptom absent) to 4 (severe symptoms).
  Scores from 0 to 82 with higher score indicating worse depression
Time Frame: Week 10
Population: subjects for whom data post baseline were available
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
scores on a scale | 19.1 (9.5) | 28.5 (14.6)
Statistical Analysis 1: Comparison: Duloxetine (Cymbalta) vs Placebo Treatment; Repeated measures ANOVA was used to compare measures between baseline and week 10; Test type: Superiority or Other; p = 0.05, Repeated Measures ANOVA; d.f. 1,55; F statistics = 8.72 — Time x Treatment: F=8.72, d.f=1,55, p=0.05

4. Secondary Outcome: Global Assessment of Functioning Scale (GAF)
Description: A commonly used rating scale for global social function.
  Range from 0 to 100; higher score=better functioning. 91 - 100 No symptoms. 81 - 90 Absent or minimal symptoms 71 - 80 no more than slight impairment in social, occupational, or school functioning (e.g., temporarily falling behind in schoolwork).
  61 - 70 Some mild symptoms 51 - 60 Moderate symptoms 41 - 50 Serious symptoms 31 - 40 Some impairment in reality testing or communication 21 - 30 Behavior is considerably influenced by delusions or hallucinations or serious impairment, in communication or judgment 11 - 20 Some danger of hurting self or others
  1 - 10 Persistent danger of severely hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death.
  0 Inadequate information
Time Frame: Week 10
Population: subjects for whom post-baseline data were available
Measure: Mean (Standard Deviation); unit: points on rating scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
points on rating scale | 69.9 (20.9) | 65.7 (14)
Statistical Analysis 1: Comparison: Duloxetine (Cymbalta) vs Placebo Treatment; Repeated measures ANOVA was used to compare measures between baseline and week 10; Test type: Superiority or Other; p = 0.025, Repeated measures ANOVA; d.f. 1,55; F statistics = 5.33

5. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Beck Depression Inventory (BDI)is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-offs are as follows:[7]
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
  Higher total scores indicate more severe depressive symptoms.
Time Frame: Week 10
Population: subjects fro whom post-baseline data was available
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
Scores on a scale | 8.5 (7) | 10.1 (6.2)
Statistical Analysis 1: Comparison: Duloxetine (Cymbalta) vs Placebo Treatment; Repeated measures ANOVA was used to compare measures between baseline and week 10; Test type: Superiority or Other; p = 0.6, Repeated measures ANOVA; d.f.=1,55; F statistics = 0.26

6. Secondary Outcome: Clinical Global Impressions Improvement(CGI-I)
Description: The Clinical Global Impression - Improvement(CGI-I) is a 7-point scale that rate patient's total improvement whether or not comparing to his/her condition at baseline.
  0 = Not assessed
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse Higher score=greatest worsening
Time Frame: 10 weeks
Population: subjects for whom post-baseline data was available
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
Scores on a scale | 2.4 (.8) | 3 (1.1)

7. Secondary Outcome: Cornell Dysthymia Rating Scale (CDRS)
Description: as for outcome 3
Time Frame: Baseline
Population: subjects for whom data post baseline were available
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
Scores on a scale | 36.9 (8.0) | 37.4 (8.0)

8. Secondary Outcome: Beck Depression Inventory (BDI)
Description: as for outcome 5
Time Frame: Baseline
Population: subjects for whom post-baseline data was available
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
Scores on a scale | 12.7 (5.8) | 15.5 (5.5)

9. Secondary Outcome: Global Assessment of Functioning Scale (GAF)
Description: as for outcome 4
Time Frame: Baseline
Population: subjects for whom post-baseline data were available
Measure: Mean (Standard Deviation); unit: points on rating scale
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 29 | 28
points on rating scale | 62.6 (5.8) | 58.3 (7.0)

10. Other Pre Specified Outcome: Resting-state Functional Connectivity Magnetic Resonance Imaging(fMRI)
Description: To use resting-state fMRI to study the effects of antidepressant therapy on default mode network (DMN) connectivity density.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of connecting nods
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 15 | 17
percentage of connecting nods | 0.21 (0.08) | 0.24 (0.06)
Statistical Analysis 1: Comparison: Duloxetine (Cymbalta) vs Placebo Treatment; Test type: Other; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = 4.0

11. Other Pre Specified Outcome: Resting-state Functional Connectivity Magnetic Resonance Imaging(fMRI)
Description: as for outcome 10
Time Frame: Follow up
Measure: Mean (Standard Deviation); unit: percentage of connecting nods
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Number analyzed (Participants) | 15 | 17
percentage of connecting nods | 0.16 (0.06) | 0.19 (0.08)
Statistical Analysis 1: Comparison: Duloxetine (Cymbalta) vs Placebo Treatment; Test type: Other; p = 0.9, t-test, 2 sided; Mean Difference (Final Values) = 0.4

ADVERSE EVENTS:
Time Frame: patients were treated in study for 22 weeks, including 10 weeks double blind medication vs placebo and 12 weeks open label treatment.
Description: All started participants were assessed for Serious Adverse Events, while only completed participants were assessed for Other Adverse Events.
Arm/Group | Duloxetine (Cymbalta) | Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 27/29 | 22/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (Cymbalta) (N=29) | Placebo Treatment (N=28)
GI upset (Gastrointestinal disorders) | 7 (7) | 9 (9)
Fatigue (General disorders) | 9 (9) | 8 (8)
Nausea (General disorders) | 6 (6) | 5 (5)
Dizziness (General disorders) | 2 (2) | 4 (4)
Decreased Sleep (General disorders) | 6 (6) | 4 (4)
Decreased Appetite (General disorders) | 8 (8) | 4 (4)
Vivid Dream (General disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less